CLINICAL TRIAL: NCT00919893
Title: Phase 3 Study of a Standardized Pollen Extract Preparation (Cernilton) in Patients With Inflammatory Chronic Prostatitis-chronic Pelvic Pain Syndrome
Brief Title: Efficacy Study of a Standardized Pollen Extract Preparation (Cernilton) to Treat Inflammatory Chronic Prostatitis-Chronic Pelvic Pain Syndrome (CP-CPPS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Strathmann AG&Co, Hamburg, Germany (Unknown); Cernelle, Ängelholm, Sweden (Unknown)
Responsible Party: Prof. Dr. Wolfgang Weidner, Clinic for Urology and Pediatric Urology, JL-University, Giessen, Germany
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4015497
Record Dates: First submitted 2009-02-10; First posted 2009-06-12 (Estimated); Results first posted 2009-06-12 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2009-06

CONDITIONS: Chronic Prostatitis; Chronic Pelvic Pain Syndrome
Keywords: chronic prostatitis symptom index; male; inflammatory; CP-CPPS; Cernilton; pelvic pain; symptoms
MeSH Terms: conditions — Pelvic Pain | interventions — cernilton

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cernilton (Active Comparator): Men with inflammatory chronic prostatitis-chronic pelvic pain syndrome (CP-CPPS)
  Interventions: Drug: Cernilton
- Placebo (Placebo Comparator): Men with inflammatory chronic prostatitis-chronic pelvic pain syndrome (CP-CPPS)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cernilton — Oral Cernilton, 2 capsules every 8 hours with the active substance consisting of 23 mg Extractum Pollens siccatum, 4 mg L-glutamate and 0.23 mg Stigmasterol per capsule for 12 weeks.
  Arms: Cernilton
Drug: Placebo — Oral placebo, 2 capsules every 8 hours with identical capsulation and weight only containing the inactive substances in proportional doses as compared with Cernilton for 12 weeks.
  Arms: Placebo

SUMMARY:
In this placebo controlled study the safety and efficacy of Cernilton, a standardized pollen extract, in men with inflammatory chronic prostatitis-chronic pelvic pain syndrome was investigated. The purpose of this study is to determine whether Cernilton is safe and effective in patients with inflammatory chronic prostatitis-chronic pelvic pain syndrome.

DETAILED DESCRIPTION:
We conducted a multicenter, randomized, double-blind, placebo-controlled trial to assess safety and efficacy of Cernilton, a standardized pollen extract, in men with inflammatory CP-CPPS (National Institutes of Health (NIH) type IIIA). Participants were randomized to Cernilton or placebo for 12 weeks and were evaluated using the National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) individual domains and total score, the number of leukocytes in post prostatic massage urine, the International Prostate Symptom Score (IPSS) and the sexuality domain of a life satisfaction questionnaire at baseline and after 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* men between 18 and 65 years
* symptoms of pelvic pain for at least 3 months during the 6 months before study entry
* a score in the pain domain of the German validated version of the NIH chronic prostatitis symptom index (NIH-CPSI) of 7 or higher
* leukocytes of 10 or more in post prostate massage urine

Exclusion Criteria:

* urinary tract infection
* acute bacterial or chronic bacterial prostatitis
* history of urethritis with discharge 4 weeks prior to study entry
* a history of epididymitis or sexually transmitted disease
* residual urine volume of more than 50 mL due to bladder outlet obstruction
* indication for or history of prostate surgery including prostate biopsy
* treatment with phytotherapeutic agents
* alpha-blocker agents or antimicrobial substances with prostatic penetration 4 weeks prior to study entry
* treatment with agents influencing intraprostatic hormone metabolism 6 months prior to study entry

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 1999-12; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Weidner, Prof. Dr., Principal Investigator — Clinic for Urology and Pediatric Urology, Justus-Liebig-University Giessen, Germany
Locations (1):
- Justus-Liebig-University, Giessen, Germany

REFERENCES:
- [Background] Rugendorff EW, Weidner W, Ebeling L, Buck AC. Results of treatment with pollen extract (Cernilton N) in chronic prostatitis and prostatodynia. Br J Urol. 1993 Apr;71(4):433-8. doi: 10.1111/j.1464-410x.1993.tb15988.x. PMID 8499988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients at urologic clinics. Start date: December 1999. Stop date: January 2004.
Groups:
- Cernilton: Oral Cernilton, 2 capsules every 8 hours with the active substance consisting of 60 mg Cernitin T60 (water-soluble fraction) and 3 mg Cernitin GBX (fat-soluble fraction)per capsule for 12 weeks.
- Placebo: Oral placebo, 2 capsules every 8 hours, identical capsulation and weight only containing the inactive substances in proportional doses as compared with Cernilton for 12 weeks.
Period: Overall Study
Arm/Group | Cernilton | Placebo
Started | 70 | 69
Completed | 51 | 60
Not Completed | 19 | 9
Not completed — Protocol Violation | 19 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cernilton | Placebo | Total
Number analyzed (Participants) | 70 | 69 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 69 | 139
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (7.2) | 39.3 (9.1) | 39.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 70 | 69 | 139
Region of Enrollment [Number; unit: participants]
  Germany | 70 | 69 | 139

OUTCOME MEASURES:

1. Secondary Outcome: Secondary Outcomes Were Symptomatic Improvement of the NIH-CPSI Total Score, the Micturition and Life Quality Domains of the NIH-CPSI Questionnaire, Decrease in the Number of Leukocytes in Urine.
Description: Decrease of score points. Decrease of leucocytes in urine.
Time Frame: 0, 6, 12 weeks
Measure: Number; unit: participants
Arm/Group | Cernilton | Placebo
Number analyzed (Participants) | 70 | 69
participants | 47 | 33

2. Primary Outcome: Symptomatic Improvement in the Pain Domain of National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI)
Description: Decrease in NIH-CPSI pain score. Best value: 0. Worst value: 21.
Time Frame: 0, 6, 12 weeks
Population: ITT (Intention to treat) LOCF (Last observation carried forward)
Measure: Number; unit: participants
Arm/Group | Cernilton | Placebo
Number analyzed (Participants) | 70 | 69
participants | 47 | 33
Statistical Analysis 1: Comparison: Cernilton vs Placebo; Null hypothesis: Cernilton compared to placebo induces a better or the same outcome of symptomatic improvement in the pain domain of symptomatic Pelvic Pain Syndrome verified by the National Institutes of Health-Chronic Prostatitis Symptom Index (NIH-CPSI). Power calculation: A power of 1-beta=0.8 was calculated; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No